CLINICAL TRIAL: NCT04068662
Title: Intervening During the Prenatal Period With Women Exposed to Intimate Partner Violence to Improve Maternal Functioning and Infant Adjustment
Brief Title: Intervention for IPV-exposed Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Collaborators: University of Memphis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-03-5260
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Postpartum Depression; Posttraumatic Stress Disorder; Infant Behavior; Violence; Parenting
Keywords: intimate partner violence; resilience, psychological
MeSH Terms: conditions — Depression, Postpartum; Stress Disorders, Post-Traumatic; Infant Behavior

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either the Pregnant Moms' Empowerment Program or an active control group. Members of the active control group participate in a non-directive support group with contact equivalent time to the Pregnant Moms' Empowerment Program (10 hrs).
Who Masked: Participant
Masking Description: All women are told that they are participating in a support group program for pregnant women who have experienced intimate partner violence, and do not receive any information about the content of either condition or their assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant Moms' Empowerment Program (Experimental): Five session group therapy program covering safety planning, resilience and coping, infant care and parenting.
  Interventions: Behavioral: Pregnant Moms' Empowerment Program
- Nondirective Support Group (Active Comparator): Five session nondirective support group with two co-leaders who assist in facilitating open discussion on women's self-identified discussion topics.
  Interventions: Behavioral: Nondirective Support Group

INTERVENTIONS:
Behavioral: Pregnant Moms' Empowerment Program — The Pregnant Moms' Empowerment Program is a five session group therapy program designed for pregnant women with a recent history of exposure to intimate partner violence. One session is administered each week with a duration of 2 hours each, for a total of ten contact hours across the course of the intervention. Intervention topics includes safety planning, social support, resilience, psychoeducation about intimate partner violence, cognitive and behavioral strategies for remediating distress, infant sleep and breastfeeding, responsive parenting, and co-parenting.
  Arms: Pregnant Moms' Empowerment Program
Behavioral: Nondirective Support Group — Participants in the non-directive support group condition participate in groups of the same size and with the same total contact time as women in Intervention 1. In contrast to the structured, manualized content delivered as a part of the Pregnant Moms' Empowerment Program, however, group leaders in this condition facilitate open conversation on topics that women identify together as a group.
  Arms: Nondirective Support Group

SUMMARY:
The overarching goal of the proposed project is to evaluate a randomized clinical trial of the Pregnant Moms' Empowerment Program aimed at detecting its effects on maternal mental health, re-victimization, parenting sensitivity, and infant development. The project also seeks to examine theoretically-grounded mechanisms of change, including social support and empowerment. Women participating in the study will receive either the PMEP or participate in a contact-equivalent active control group during pregnancy, and will be interviewed at baseline, post-intervention and with their infants at 3 months and 1 year old. The study will occur at two sites - the University of Notre Dame and the University of Memphis. Participants will be recruited from the local community at both locations, with an equal number of women drawn from each site - Memphis, Tennessee (n=115) and South Bend, Indiana (n=115). Enrollment will continue for approximately 2.5 years, with an expected rate of 8 eligible women per month, based on a pilot study of the Pregnant Moms' Empowerment Program. The expected duration of the study for each participant will be approximately 1.5 years, with some variation due to women enrolling at different points in their pregnancy.

The primary objective of the proposed project is to determine if the Pregnant Moms' Empowerment Program has positive effects on maternal mental health, re-victimization rates, parenting sensitivity, and infant development compared to women's participation in a contact-equivalent active control group. This objective will be evaluated using a multi-site randomized clinical trial design. Participants (N = 230) will be equally randomized into study arms. Eligible women will include those who are: 1) currently pregnant (primi or multiparous) and between 10 and 30 weeks gestation, 2) experienced IPV within the past year, 3) English speaking and 4) age 16 or older.

The study will include 9 total visits: 4 assessments and 5 sessions for both study arms. In-person assessment visits will be completed by a trained research assistant; each visit will take approximately 2-3 hours, with post-partum assessments somewhat longer than prenatal assessments given the addition of the infant developmental assessment and parent-child observation task. Women will be compensated $30 for the first two assessments and $50 for the second two assessments. Following the final assessment, women will be invited to complete a daily diary (virtually) each day for 30 days. Each survey will take approximately 5-10 minutes to complete, and women will be compensated $2 for each completed survey. Women will also receive a $10 bonus for each set of 10 consecutive surveys. Treatment sessions will be 2 hours in duration. Women in the PMEP will complete a structured set of sessions: (1) supporting each other, support in the community, (2) identifying and understanding sources of distress, (3) cognitive and behavioral strategies to build resilience and resolve conflict, (4) perinatal health and infant care, and (5) positive parenting. Women in the active control condition will participate in facilitated discussions on a topic identified by the group. All sessions will be audio recorded so that treatment fidelity can be evaluated (for the Pregnant Moms' Empowerment Program) and so that content overlap can be assessed (for the active control condition).

DETAILED DESCRIPTION:
The study will occur at two sites - the University of Notre Dame and the University of Memphis. Participants will be recruited from the local community at both locations, with an equal number of women drawn from each site (n=115 at each site for a total of N=230 mothers). Enrollment will continue for approximately 2.5 years, with an expected rate of 8 eligible women per month, based on a pilot study of the PMEP. The expected duration of the study for each participant is approximately 1.75 years, with some variation due to women enrolling at different points in their pregnancy. The primary objective of the current study is to determine if the PMEP has positive effects on maternal mental health, re-victimization rates, parenting sensitivity, and infant development, as compared to women's participation in a contact-equivalent control group. This objective will be evaluated usin ga multi-site randomized clinical trial design. Participants (N=230) will be equally randomized into study arms. Eligible women include those who are currently pregnant, who have experienced IPV in the past year, are age 16 or older, and are currently between 10 and 30 weeks pregnant. In-person assessment visits will be completed by a trained research assistant; each visit will take approximately 2-3 hours, with postpartum assessments somewhat longer than prenatal assessments due to the addition of the infant developmental assessment. Women will be compensated $30 for the first two assessments and $50 for the second two assessments. Treatment sessions will be 2 hrs in duration. Women in the PMEP will complete a structured set of sessions: (1) safety planning, (2) identifying and understanding sources of distress, (3) cognitive and behavioral strategies to build resilience and resolve conflict, (4) perinatal health and infant care, (5) positive parenting. Women in the AC will participate in facilitated discussions on a topic identified by the group. All sessions will be audiorecorded so that treatment fidelity can be evaluated (for PMEP) and content overlap can be identified (for AC).

ELIGIBILITY:
Inclusion Criteria:

* currently pregnant (primi or multiparous)
* experienced intimate partner violence within the past year
* English speaking
* age 16 or older
* between 10-30 weeks pregnant

Exclusion Criteria:

* fails to meet inclusion criteria
* unavailable or unwilling to participate in core study components, including groups

Ages: 3 Months to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 424 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Change in posttraumatic stress symptoms from baseline to post-treatment | posttreatment
  Mothers will report on symptoms of posttraumatic stress using the PTSD Checklist for DSM-5 (Weathers, Litz, Keane, Palmieri, Marx, & Schnurr, 2013). We hypothesize that compared to women in the active control condition, that beginning at the post-treatment assessment women in the treatment condition will have lower levels of posttraumatic stress. Further, we hypothesize that this will be mediated by the effect of treatment on women's empowerment and social support. Items are summed to create a total score, which can range from 0 to 80. Higher scores indicate worse outcomes.
Change in posttraumatic stress symptoms from baseline to 3-months postpartum | 3-months postpartum
  Mothers will report on symptoms of posttraumatic stress using the PTSD Checklist for DSM-5 (Weathers, Litz, Keane, Palmieri, Marx, & Schnurr, 2013). We hypothesize that compared to women in the active control condition, women in the treatment condition will have lower levels of posttraumatic stress. Further, we hypothesize that this will be mediated by the effect of treatment on women's empowerment and social support. Items are summed to create a total score, which can range from 0 to 80. Higher scores indicate worse outcomes.
Change in posttraumatic stress symptoms from baseline to 12-months postpartum | 12-months postpartum
  Mothers will report on symptoms of posttraumatic stress using the PTSD Checklist for DSM-5 (Weathers, Litz, Keane, Palmieri, Marx, & Schnurr, 2013). We hypothesize that compared to women in the active control condition, women in the treatment condition will have lower levels of posttraumatic stress. Further, we hypothesize that this will be mediated by the effect of treatment on women's empowerment and social support. Items are summed to create a total score, which can range from 0 to 80. Higher scores indicate worse outcomes.
Change in depressed mood from baseline to posttreatment | posttreatment
  Mothers will report on symptoms of depressed mood using the Center for Epidemiological Studies Depression Scale (Radloff, 1977). We hypothesize that compared to women in the AC condition, that beginning at the post-treatment assessment (T2) women in the PMEP condition will have lower levels of depressed mood over time. Further, we hypothesize that this will be mediated by the effect of treatment on women's empowerment and social support. Items are summed to create a total score, which can range from 0 to 60. Higher scores indicate worse outcomes.
Change in depressed mood from baseline to 3-months postpartum | 3-months postpartum
  Mothers will report on symptoms of depressed mood using the Center for Epidemiological Studies Depression Scale (Radloff, 1977). We hypothesize that compared to women in the active control condition, that beginning at that women in the treatment condition will have lower levels of depressed mood over time. Further, we hypothesize that this will be mediated by the effect of treatment on women's empowerment and social support. Items are summed to create a total score, which can range from 0 to 60. Higher scores indicate worse outcomes.
Change in depressed mood from baseline to 12-months postpartum | 12-months postpartum
  Mothers will report on symptoms of depressed mood using the Center for Epidemiological Studies Depression Scale (Radloff, 1977). We hypothesize that compared to women in the active control condition, that beginning at that women in the treatment condition will have lower levels of depressed mood over time. Further, we hypothesize that this will be mediated by the effect of treatment on women's empowerment and social support. Items are summed to create a total score, which can range from 0 to 60. Higher scores indicate worse outcomes.
Change in resilience from baseline to posttreatment | posttreatment
  Mothers will report on resilience using the Connor-Davidson Resilience Scale (Connor & Davidson, 2003), which examines one's ability to cope with adversity. We hypothesize that compared to women in the active control condition that women in the treatment condition will have higher levels of resilience over time. Further, we hypothesize that this will be mediated by the effect of treatment on women's empowerment and social support. Items are summed to create a total score, which can range from 0 to 100. Higher scores indicate better outcomes.
Change in resilience from baseline to 3-months postpartum | 3-months postpartum
  Mothers will report on resilience using the Connor-Davidson Resilience Scale (Connor & Davidson, 2003), which examines one's ability to cope with adversity. We hypothesize that compared to women in the active control condition that women in the treatment condition will have higher levels of resilience over time. Further, we hypothesize that this will be mediated by the effect of treatment on women's empowerment and social support. Items are summed to create a total score, which can range from 0 to 100. Higher scores indicate better outcomes.
Change in resilience from baseline to 12-months postpartum | 12-months postpartum
  Mothers will report on resilience using the Connor-Davidson Resilience Scale (Connor & Davidson, 2003), which examines one's ability to cope with adversity. We hypothesize that compared to women in the active control condition that women in the treatment condition will have higher levels of resilience over time. Further, we hypothesize that this will be mediated by the effect of treatment on women's empowerment and social support. Items are summed to create a total score, which can range from 0 to 100. Higher scores indicate better outcomes.
Maternal Sensitivity at infant age 3 months | 3-months postpartum
  Maternal sensitivity will be assessed using observational paradigms coded by trained research assistants for sensitive parenting behaviors. At the 3 month and 12 month postpartum assessments, mother-infant dyads will participate in a fixed-order observational assessment, constituted of the Still-Face Paradigm (Tronick et al., 1978) and a 10-minute free play period. Parent sensitivity will be rated on a 5 point Likert scale from the play and reunion episodes. Coded ratings on sensitivity and intrusiveness will be combined across intervals to create a composite maternal sensitivity score. We hypothesize that compared to women in the active control condition, women in the treatment condition will show higher levels of maternal sensitivity at the 3-month postpartum assessment. Higher scores indicate better outcomes.
Maternal Sensitivity at infant age 12 months | 12-months postpartum
  Maternal sensitivity will be assessed using observational paradigms coded by trained research assistants for sensitive parenting behaviors. At the 3 month and 12 month postpartum assessments, mother-infant dyads will participate in a fixed-order observational assessment, constituted of the Still-Face Paradigm (Tronick et al., 1978) and a 10-minute free play period. Parent sensitivity will be rated on a 5 point Likert scale from the play and reunion episodes. Coded ratings on sensitivity and intrusiveness will be combined across intervals to create a composite maternal sensitivity score. We hypothesize that compared to women in the active control condition, women in the treatment condition will show higher levels of maternal sensitivity at the 12-month postpartum assessment. Higher scores indicate better outcomes.
Intimate Partner Violence at posttreatment | posttreatment
  The Revised Conflict Tactics Scale (Straus, et al, 1996) will be used to assess the severity of psychological, physical, and sexual violence experienced by women in a dating, cohabiting, or marital relationship. We hypothesize that compared to women in the active control condition that women in the treatment condition will have lower frequency of intimate partner re-victimization over time. Further, we hypothesize that this will be mediated by the effect of treatment on women's empowerment and social support. Items cluster into five scales: physical assaults, psychological aggression, sexual coercion, injury, and negotiation techniques. Respondents report frequency on a scale of 1 = once [since the last interview] to 6 = more than 20 times [since the last interview]. Higher scores indicate worse outcomes. The current study used the frequency scoring method for the CTS2, which recodes the scale to represent the midpoints of each range with a possible total range of 0 to 825 events.
Intimate Partner Violence at 3-months postpartum | 3-months postpartum
  he Revised Conflict Tactics Scale (Straus, et al, 1996) will be used to assess the severity of psychological, physical, and sexual violence experienced by women in a dating, cohabiting, or marital relationship. We hypothesize that compared to women in the active control condition that women in the treatment condition will have lower frequency of intimate partner re-victimization over time. Further, we hypothesize that this will be mediated by the effect of treatment on women's empowerment and social support. Items cluster into five scales: physical assaults, psychological aggression, sexual coercion, injury, and negotiation techniques. Respondents report frequency on a scale of 1 = once [since the last interview] to 6 = more than 20 times [since the last interview]. Higher scores indicate worse outcomes. The current study used the frequency scoring method for the CTS2, which recodes the scale to represent the midpoints of each range with a possible total range of 0 to 825 events.
Intimate Partner Violence at 12-months postpartum | 12-months postpartum
  he Revised Conflict Tactics Scale (Straus, et al, 1996) will be used to assess the severity of psychological, physical, and sexual violence experienced by women in a dating, cohabiting, or marital relationship. We hypothesize that compared to women in the active control condition that women in the treatment condition will have lower frequency of intimate partner re-victimization over time. Further, we hypothesize that this will be mediated by the effect of treatment on women's empowerment and social support. Items cluster into five scales: physical assaults, psychological aggression, sexual coercion, injury, and negotiation techniques. Respondents report frequency on a scale of 1 = once [since the last interview] to 6 = more than 20 times [since the last interview]. Higher scores indicate worse outcomes. The current study used the frequency scoring method for the CTS2, which recodes the scale to represent the midpoints of each range with a possible total range of 0 to 825 events.
Infant Development at 3 months of age | 3-months
  Infant development (cognitive, language, socioemotional) will be evaluated using The Bayley Scales of Infant and Toddler Development and The Ages and Stages Questionnaire - 3, which are a standardized measures. We hypothesize that compared to infants born to women in the active control condition, infants born to mothers in the treatment condition will show better developmental outcomes. Further, we hypothesize that infant development at 12 months will be indirectly predicted by mothers' improvement as a result of treatment at 3 months. The Bayley is a standardized measure and within each domain an average score is 100. Higher scores indicate better outcomes. On the Ages and Stages Questionnaire, scores for each subdomain (Communication, Gross Motor, Fine Motor, Problem Solving, and Personal-Social) range from 0 to 60.
Infant Development at 12 months of age | 12-months
  Infant development (cognitive, language, socioemotional) will be evaluated using The Bayley Scales of Infant and Toddler Development and The Ages and Stages Questionnaire - 3, which are a standardized measures. We hypothesize that compared to infants born to women in the active control condition, infants born to mothers in the treatment condition will show better developmental outcomes. Further, we hypothesize that infant development at 12 months will be indirectly predicted by mothers' improvement as a result of treatment at 3 months. The Bayley is a standardized measure and within each domain an average score is 100. Higher scores indicate better outcomes. On the Ages and Stages Questionnaire, scores for each subdomain (Communication, Gross Motor, Fine Motor, Problem Solving, and Personal-Social) range from 0 to 60.
Infant Regulation at 3 months of age | 3-months
  At the 3 month and 12 month postpartum assessments, mother-infant dyads will participate in the Still-Face Paradigm (Tronick et al., 1978). Infant affect, which includes a combination of vocal and facial reactions, will be rated on a second-by-second basis across all three episodes of the SFP and free play. A 7 point Likert scale ranging from a -3 (screaming) to +3 (laughing intensely) will be used. Affect data are reduced to the proportion of time infants spend in negative and positive affect states (Braungart-Rieker et al., 2014). We hypothesize that compared to infants born to women in the active control condition, infants born to mothers in the treatment condition will show more positive affect over time, at 3 and 12 months of age. Further, we hypothesize that infant affect at 12 months will be indirectly predicted by mothers' improvement as a result of treatment at 3 months. Higher scores indicate better outcomes.
Infant Regulation at 12 months of age | 12-months
  At the 3 month and 12 month postpartum assessments, mother-infant dyads will participate in the Still-Face Paradigm (Tronick et al., 1978). Infant affect, which includes a combination of vocal and facial reactions, will be rated on a second-by-second basis across all three episodes of the SFP and free play. A 7 point Likert scale ranging from a -3 (screaming) to +3 (laughing intensely) will be used. Affect data are reduced to the proportion of time infants spend in negative and positive affect states (Braungart-Rieker et al., 2014). We hypothesize that compared to infants born to women in the active control condition, infants born to mothers in the treatment condition will show more positive affect over time, at 3 and 12 months of age. Further, we hypothesize that infant affect at 12 months will be indirectly predicted by mothers' improvement as a result of treatment at 3 months. Higher scores indicate better outcomes.

SECONDARY OUTCOMES:
Change in social support from baseline to posttreatment | posttreatment
  Women's sources of maternal support will be assessed with the Lubben Social Network Scale-Revised(Lubben & Gironda, 2003), which examines the level of perceived support from family networks and friendship networks. We hypothesize that compared to women in the active control condition, that women in the treatment condition will have higher social support over time. Further, we hypothesize that social support will mediate the relationship between treatment and women's mental health, revictimization, resilience, and sensitive parenting. Total scores range from 0 to 90. Higher scores indicate better outcomes.
Change in social support from baseline to 3-months postpartum | 3-months postpartum
  Women's sources of maternal support will be assessed with the Lubben Social Network Scale-Revised(Lubben & Gironda, 2003), which examines the level of perceived support from family networks and friendship networks. We hypothesize that compared to women in the active control condition, that women in the treatment condition will have higher social support over time. Further, we hypothesize that social support will mediate the relationship between treatment and women's mental health, revictimization, resilience, and sensitive parenting. Total scores range from 0 to 90. Higher scores indicate better outcomes.
Change in social support from baseline to 12-months postpartum | 12-months postpartum
  Women's sources of maternal support will be assessed with the Lubben Social Network Scale-Revised(Lubben & Gironda, 2003), which examines the level of perceived support from family networks and friendship networks. We hypothesize that compared to women in the active control condition, that women in the treatment condition will have higher social support over time. Further, we hypothesize that social support will mediate the relationship between treatment and women's mental health, revictimization, resilience, and sensitive parenting. Total scores range from 0 to 90. Higher scores indicate better outcomes.
Change in empowerment from baseline to posttreatment | posttreatment
  The Personal Progress Scale-Revised (Johnson, Worrell, & Chandler, 2005) will be used to examine women's attitudes and behaviors associated with increased empowerment and well-being. We hypothesize that compared to women in the active control condition, that women in the treatment condition will have higher empowerment over time. Further, we hypothesize that empowerment will mediate the relationship between treatment and women's mental health, revictimization, resilience, and sensitive parenting. Scores range from 0 to 196; higher scores indicated better outcomes.
Change in empowerment from baseline to 3-months postpartum | 3-months postpartum
  The Personal Progress Scale-Revised (Johnson, Worrell, & Chandler, 2005) will be used to examine women's attitudes and behaviors associated with increased empowerment and well-being. We hypothesize that compared to women in the active control condition, that women in the treatment condition will have higher empowerment over time. Further, we hypothesize that empowerment will mediate the relationship between treatment and women's mental health, revictimization, resilience, and sensitive parenting. Scores range from 0 to 196; higher scores indicated better outcomes.
Change in empowerment from baseline to 12-months postpartum | 12-months postpartum
  The Personal Progress Scale-Revised (Johnson, Worrell, & Chandler, 2005) will be used to examine women's attitudes and behaviors associated with increased empowerment and well-being. We hypothesize that compared to women in the active control condition, that women in the treatment condition will have higher empowerment over time. Further, we hypothesize that empowerment will mediate the relationship between treatment and women's mental health, revictimization, resilience, and sensitive parenting. Scores range from 0 to 196; higher scores indicated better outcomes.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Notre Dame, Notre Dame, Indiana
  - University of Memphis, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Five years after the completion of the study we will make the data available to other researchers for the purposes of replication of published findings or inclusion of data in meta-analyses via a data-sharing agreement that will provide for: (1) a commitment to using the data only for these research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available for five years after the completion of the study.
Access Criteria: Interested persons will contact PIs Miller-Graff and Howell to arrange a datasharing agreement

DOCUMENTS (1):
  • Informed Consent Form (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT04068662/ICF_001.pdf